CLINICAL TRIAL: NCT07027657
Title: Safety and Efficacy of BTL-699-2 for the Improvement of Sleep Quality and Reduction of Stress
Brief Title: EXOMIND (BTL-699-2) for the Improvement of Sleep Quality and Reduction of Stress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BTL-699_CTUS300
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-07-21 (Actual); Status verified 2025-07

CONDITIONS: Sleep Quality; Stress Reduction
Keywords: rTMS; TMS; Sleep Quality; Stress Reduction; ExoTMS; EXOMIND
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: All patients will be randomly divided into 2 study groups - Group A and Group B (sham). The allocation of subjects into study groups will be in ratio 3:1 (Group A:Group B).
Who Masked: Participant
Masking Description: Only the subject will be unaware of the group assignment. The operator providing the treatment will be aware of the subject's group assignment and will perform the treatment with the setting according to the subject's group.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A - active (Active Comparator): Group A will receive transcranial magnetic stimulation treatment with the intensity of up to 70% of their motor treshold with the BTL-699-2 device.
  Interventions: Device: Treatment with BTL-699-2
- Group B - sham (Sham Comparator): Group B will receive transcranial magnetic stimulation treatment with the intensity of 5% of their motor treshold with the BTL-699-2 device.
  Interventions: Device: Treatment with BTL-699-2 (sham)

INTERVENTIONS:
Device: Treatment with BTL-699-2 — Six transcranial magnetic stimulation treatments with the BTL-699-2 device will be delivered over the left dorsolateral prefrontal cortex, spaced 3 to 7 days apart. The intensity will be adjusted according to the subject's feedback, up to 70% of the individual's motor threshold.
  Other Names: ExoTMS; EXOMIND
  Arms: Group A - active
Device: Treatment with BTL-699-2 (sham) — Six transcranial magnetic stimulation treatments with the BTL-699-2 device will be delivered over the left dorsolateral prefrontal cortex, spaced 3 to 7 days apart. The intensity will be adjusted according to the subject's feedback, up to 5% of the individual's motor threshold.
  Other Names: ExoTMS; EXOMIND
  Arms: Group B - sham

SUMMARY:
The goal of this clinical trial is to evaluate whether the treatment with BTL-699-2 device is able to improve sleep quality and reduce stress in adults above the age of 22 years. The main questions it aims to answer are:

Does the treatment with BTL-699-2 device improve sleep quality? Does the treatment with BTL-699-2 device reduce stress?

Participants will be asked to:

* Undergo six treatments
* Complete the Pittsburgh Sleep Quality Index
* Complete the Perceived Stress Scale Questionnaire
* Complete the Sleep and Stress Assessment Questionnaire
* Complete the Therapy Comfort and Subject Satisfaction Questionnaire

DETAILED DESCRIPTION:
The study uses a multi-center, sham-controlled, single-blinded, interventional study design. The subjects will be enrolled and assigned to two experimental study arms - Group A and Group B in the ratio 3:1. Group A will receive active treatment and Group B, which received sham treatment, will serve as a control. All enrolled participants will receive six treatment visits, 3-7 days apart.

The Pittsburgh Sleep Quality Index, Perceived Stress Scale Questionnaire and Sleep and Stress Assessment Questionnaire will be administered to the subjects before the first treatment, after the last treatment, and at the two follow-up visits - 1 month and 3 months after the final session.

The Therapy Comfort Questionnaire will be administered after the last treatment, while the Subject Satisfaction will be given after the last treatment and at both follow-up visits.

The total expected duration of subject participation, from the baseline visit to study completion, is approximately five months.

ELIGIBILITY:
Inclusion Criteria:

* Age > 22 years
* The minimal pre-treatment PSQI score of >= 5 points
* Ability to determine the motor threshold of the participant. The participant's motor threshold could be established as the minimum stimulus required to induce contraction of the right thumb
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure for the improvement in sleep quality and reduction of stress, including non-invasive brain stimulation treatments other than the study procedure during study participation
* Subjects willing and able to maintain their regular (pre-procedure) diet and exercise regimen without affecting significant change in either direction during study participation
* Willingness to comply with study instructions and to return to the clinic for the required visits
* Women of child-bearing potential* are required to use birth control measures during the whole duration of the study
* If applicable, subjects will be maintained on pre-study prescribed medications at a stable therapeutic dosage for at least 2 months prior to study entry
* Subject is not using any sleeping medication or is using over-the-counter pills (except Valerian and St. John's Wort) no more than 4 times a week

Exclusion Criteria:

* Electronic implants in or near the head - rTMS devices are contraindicated for use in patients who have active or inactive implants in or near the head including device leads, deep brain stimulators, cochlear implants, ocular implants, and vagus nerve stimulators, implanted devices such as cardiac pacemakers, defibrillators, and neurostimulators
* Metallic, ferromagnetic or other magnetic-sensitive implants/objects in or near the head - rTMS devices are contraindicated for use in patients who have conductive, ferromagnetic or other magnetic-sensitive metals implanted in their head (with some exceptions in the mouth - see Operator's Manual) or within 12 in (30 cm) of the therapy coil. (Examples include implanted electrodes/stimulators, aneurysm clips or coils, stents, bullet fragments, jewelry, hair barrettes and tattoos with metallic ink),
* Drug pumps (within 12 in (30 cm) of the therapy coil)
* Application in the heart area
* Persons with a tendency to seizure (hypotonic, epileptic)
* Ongoing anticoagulation therapy
* Ongoing severe or life-threatening condition
* Pulmonary insufficiency
* Heart disorders
* Renal insufficiency
* Decompensated* hemorrhagic conditions, blood coagulation disorders, cardiovascular diseases
* Malignant tumor, benign tumor
* Fever
* Ongoing pregnancy
* Suicidal tendencies or recent attempt to commit suicide
* Concurrent use of electroconvulsive therapy or vagus nerve stimulation
* Substance-induced depression or depression secondary to a general medical condition
* Seasonal affective disorder
* Substance abuse, obsessive compulsive disorder or post-traumatic stress disorder, major depression
* Psychotic disorder including schizoaffective disorder, bipolar disease or major depression with psychotic features
* Neurological disorders, including a history of seizures, cerebrovascular disease, primary or secondary tumors in CNS, cerebral aneurysm, dementia or movement disorders
* History of increased intracranial pressure or head trauma
* Nursing
* Usage of prescription sleep medication, Valerian of St. John's Wort in the past 2 months
* Usage of over-the-counter pills 5 or more times a week

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-02 (Actual); Primary Completion 2025-11-02 (Estimated); Study Completion 2026-08-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of Sleep Quality Improvement | 15 months
  The change in the score obtained from the Pittsburgh Sleep Quality Index will be recorded. The questionnaire will be administered at the baseline visit, after the last treatment, at the 1-month and 3-month follow-up visits. It is a 19-item questionnaire. These 19 questions are grouped into 7 components, and each component is scored on a 0 - 3 scale. The minimum obtained score is 0 and the maximum is 21. Lower score indicates healthier sleep quality, therefore improvement is considered a decrease in the obtained score.

SECONDARY OUTCOMES:
Assessment of Stress | 15 months
  Evaluation of a change in the score obtained from the Perceived Stress Scale for the assessment of the stress reduction potential. The questionnaire will be administered at the baseline visit, after the last treatment, at the 1-month and 3-month follow-up visits. Each question is rated on a 0 - 4 scale, where 0 = never, and 4 = very often. The minimum obtained score is 0 and the maximum is 40. Higher scores indicate higher levels of perceived stress.
Sleep and Stress Assessment Questionnaire | 15 months
  Sleep and Stress Assessment Questionnaire is a self-report questionnaire used to provide more insight into sleep and stress medication use and stress levels. Subjects will be asked to fill in the questionnaire at the baseline visit, after the last treatment, at 1-month and 3-month follow-up visits. The baseline questionnaire consists of 5 items, while the versions administered after the last treatment and at follow-up visits contain 6 items. The questionnaire is not scored; instead, it includes yes/no and open-ended questions to capture qualitative information on sleep and stress-related factors.
Assessment of Therapy Comfort | 15 months
  Therapy Comfort questionnaire will be used for evaluating the comfort during the treatment sessions. The Therapy Comfort questionnaire will be administered after the last treatment. Therapy Comfort questionnaire consists of the question "I found the treatment comfortable", to which responses are based on a 5-point Likert scale (1 = "strongly disagree", and 5 = "strongly agree") and the 10-point Numeric Analog Scale for pain (0 = "no pain", 10 = "worst possible pain"). A higher score for the statement "I found the treatment comfortable", and lower score on the Numeric Analog Scale for pain indicate higher therapy comfort.
Assessment of Satisfaction | 15 months
  Subject Satisfaction with treatment outcomes will be assessed using 5-point Likert Scale Subjects Satisfaction. The questionnaire will be administered after the last treatment, at the 1-month and 3-month follow-up visits. Responses to questions about satisfaction with the treatment outcomes will range from "strongly disagree" (1 point) to "strongly agree" (5 points). A higher score for each statement indicate better outcomes.
Incidence of Treatment-related Adverse Events | 15 months
  Monitoring of adverse reactions and side effects will be performed for the evaluation of safety of the treatment with the BTL-699-2 device for the improvement of sleep and reduction of stress and to identify side effects and adverse events associated with the study treatment.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - AntiAging and Wellness, Chula Vista, California
  - Kind Health Group, Encinitas, California
  - Minooka Healthcare Center, Minooka, Illinois